CLINICAL TRIAL: NCT03566927
Title: FLEX®-DCB Dialysis ACCESS Stenosis Study
Acronym: AVAFLEX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to warning letters issued regarding paclitaxel
Sponsor: VentureMed Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLEX-DCB 0518-2
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Arteriovenous Fistula
Keywords: Arteriovenous Fistula; Vascular Fistula; Scoring; Fistula; Cardiovascular Disease
MeSH Terms: conditions — Arteriovenous Fistula; Vascular Fistula; Fistula; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- FLEX Scoring Catheter plus DCB (Experimental): This is a single-arm study. All patients will be treated with the FLEX Scoring Catheter, then a standard balloon angioplasty, followed by a Lutonix® drug-coated balloon (DCB).
  Interventions: Combination Product: FLEX Scoring Catheter with Lutonix DCB

INTERVENTIONS:
Combination Product: FLEX Scoring Catheter with Lutonix DCB — Treatment by the FLEX Scoring Catheter, a plain balloon angioplasty, followed by a Lutonix DCB.

SUMMARY:
This prospective, single arm, single-center study is designed to evaluate the performance of the FLEX Scoring Catheter®/POBA/DCB in A-V access circuits.

ELIGIBILITY:
Inclusion Criteria:

* Patient is legally competent, has been informed of the study, voluntarily agrees to participate, and has signed the informed consent form.
* Arteriovenous fistula is located in the arm.
* Native AV fistula / graft was created ≥ 30 days prior to the initial procedure and has undergone at least one hemodialysis sessions.
* Venous stenosis of the AV fistula / graft with the target lesion located from the anastomosis to the axillosubclavian junction and an abnormality attributable to the stenosis as defined by K/DOQI guidelines.
* Patients with a dysfunctional or thrombosed hemodialysis access and a >50% stenosis, regardless of prior treatment (All types of lesion and access failure)
* If AV access is thrombosed, must undergo a successful thrombectomy with minimal residual thrombus.
* Intended target lesion or if a tandem lesion can be treated with ≤120 mm of DCBs in length.

Exclusion Criteria:

* Life expectancy < 9 months
* Women who are pregnant, lactating, or planning on becoming pregnant during the duration of the study.
* The hemodialysis access is located in the leg.
* Patient has more than two lesions in the access circuit.
* Patient has a secondary non-target lesion that cannot be successfully treated
* Target lesion is located central to the axillosubclavian junction.
* Surgical revision of the access site planned.
* Recent surgical interventions of the access site.
* Known allergy or sensitivity to iodinated contrast media, that cannot be adequately managed with pre- and post-procedure medication.
* Known allergy or sensitivity to paclitaxel.
* Patients who are taking immunosuppressive therapy, or routinely taking ≥ 10 mg of prednisone per day.
* Patients who have a medical condition, in the opinion of the Investigator, that may cause the patient to be noncompliant to the protocol or confound the data.
* Patients anticipating a kidney transplant.
* Patients anticipating a conversion to peritoneal dialysis.
* The patient has a stent located in the target or secondary non-target lesion.
* Patient has an active infection in the AV access or a systemic infection.
* Known hyper-coagulable state
* Currently participating in an investigational drug, biologic, or device study.
* Previously enrolled in this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Target Lesion Primary Patency | 9 Months
  Target Lesion Primary Patency at 9 months defined as the time interval of uninterrupted patency from initial study treatment to the next access thrombosis or intervention performed on the target lesion.

SECONDARY OUTCOMES:
Index of Patency Function | 3, 6, 9 Months
  Index of Patency Function defined as the average time between interventions.
Assess Secondary Patency | 3, 6, 9 Months
  Assess Secondary Patency defined as the time interval from initial study treatment to abandonment of the vascular access circuit.
Number of Interventions | 9 Months
  Mean cumulative interventions per subjects over study duration.
Percentage of Patients with Freedom from Adverse Events | 1 Month
  Freedom from major device, procedure and treatment site-related adverse events through 30 days' post procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Dialysis Access Institute, Orangeburg, South Carolina, United States